CLINICAL TRIAL: NCT07212569
Title: Analysis of Differences in Small Intestinal Microbiota Structure and Metabolites Between Patients With Irritable Bowel Syndrome and Healthy Individuals
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: xmzsyyky-2025-137
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; small intestinal microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: All participants ingest an intestinal sampling capsule for small intestinal fluid collection. Upon capsule retrieval, the samples are analyzed for their microbial DNA and metabolite content.
- Control Group: All participants ingest an intestinal sampling capsule for small intestinal fluid collection. Upon capsule retrieval, the samples are analyzed for their microbial DNA and metabolite content.

SUMMARY:
Irritable Bowel Syndrome (IBS) is a common functional bowel disorder with complex and not yet fully elucidated pathophysiological mechanisms. Recent research suggests that gut microbiota dysbiosis, particularly small intestinal bacterial overgrowth (SIBO), may play a key role in the generation of IBS symptoms. However, the vast majority of current studies have focused on fecal samples, which primarily reflect the colonic microbiota. The small intestinal microbiota, which is directly involved in nutrient digestion and absorption and more prone to dysbiosis, remains understudied due to the challenges in obtaining samples.

DETAILED DESCRIPTION:
This study aims to utilize intestinal sampling capsules to directly collect small intestinal fluid samples from both IBS patients and healthy controls. The community structure, diversity, and compositional differences of the small intestinal microbiota will be analyzed using 16S rRNA gene sequencing and metagenomic sequencing technologies, while the metabolic profiles of the small intestinal fluid will be detected via untargeted metabolomics.

ELIGIBILITY:
Inclusion Criteria:

Experimental Group： Aged 18-65 years, male or female. Meets the Rome IV diagnostic criteria for IBS The absence of organic gastrointestinal disease that could explain the symptoms.

Provides informed consent and voluntarily signs the informed consent form. Control Group： Age and sex-matched to the IBS patient group. No history of chronic digestive diseases or current gastrointestinal symptoms. Has not used antibiotics, proton pump inhibitors, probiotics, or other medications known to affect gut microbiota within the past month.

Provides informed consent and voluntarily signs the informed consent form.

Exclusion Criteria:

History of gastrointestinal surgery (excluding appendectomy). Presence of concomitant organic gastrointestinal diseases (e.g., inflammatory bowel disease, celiac disease, gastrointestinal tumors).

Presence of severe concomitant cardiac, hepatic, renal, endocrine, hematologic, or neurological diseases.

Long-term use of medications known to affect gastrointestinal motility (e.g., opioids).

Pregnancy, lactation, or women planning a pregnancy. Conditions contraindicating the use of capsule endoscopy, such as dysphagia, or known gastrointestinal strictures, diverticula, or obstruction.

Any other condition deemed by the investigator as unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort included Rome IV-diagnosed IBS patients without confounding surgical or medication history, along with age- and sex-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Identify the specific differences in the core architecture of the small intestinal microbiota between IBS patients and healthy individuals. | 6 Months
  Intestinal content samples from different regions were collected from IBS patients and healthy subjects using smart enteric-coated sampling capsules. These samples subsequently underwent 16S rRNA gene sequencing and metagenomic sequencing to analyze microbial composition, alongside untargeted metabolomics to detect metabolic differences. The regional variations in both the microbiome and metabolome were then analyzed in the IBS cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- Hongzhi Xu, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No